CLINICAL TRIAL: NCT01354171
Title: Active Surveillance Magnetic Resonance Imaging Study
Acronym: ASIST
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Canadian Urology Research Consortium (Other)
Collaborators: Ontario Institute for Cancer Research (Other); Eigen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CURC-003
Record Dates: First submitted 2011-05-13; First posted 2011-05-16 (Estimated); Last update posted 2016-10-14 (Estimated); Status verified 2012-03

CONDITIONS: Prostate Cancer
Keywords: active surveillance; low risk prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TRUS guided biopsy (No Intervention)
- MRI Assisted TRUS guided biopsy (Experimental)
  Interventions: Device: MRI assisted TRUS guided biopsy

INTERVENTIONS:
Device: MRI assisted TRUS guided biopsy — All subjects to have a confirmatory biopsy at one year. Those assigned ARM 1 to have a TRUS guided biopsy and those assigned to ARM 2to have a MRI assisted TRUS guided biopsy
  Arms: MRI Assisted TRUS guided biopsy

SUMMARY:
This is a multi-centre, prospective, randomized phase III trial to determine if multi-parametric Magnetic Resonance Imaging (MRI) can improve selection of patients eligible for active surveillance through better detection of clinically significant cancer.

ELIGIBILITY:
Inclusion Criteria:

* histological confirmation of adenocarcinoma of the prostate
* candidate for active surveillance (favourable risk prostate cancer) as defined by the following:

  * Clinical stage T1b, T1c, T2a or T2b at the time of diagnosis
  * Clinical (diagnostic biopsy) Gleason sum < 6
  * PSA < 10.0 ng/ml (ug/L)

Exclusion Criteria:

* Previous treatment for prostate cancer including surgery (excluding biopsy), radiation therapy, hormonal therapy (e.g. megestrol, medroxyprogesterone, cyproterone, DES), glucocorticoids (except inhaled or topical), LHRH analogues (e.g. Leuprolide, goserelin), ketoconazole, non-steroidal antiandrogens (e.g. bicalutamide, flutamide) and/or any 5α-reductase inhibitors within 3 months of randomization
* Planned anti-androgen therapy
* Inability to undergo TRUS biopsy
* Inability to undergo multi-parametric MRI

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2011-11; Primary Completion 2016-09 (Actual); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
To determine the proportion of subjects whose confirmatory biopsy is upgraded to Gleason score 7 (3+4) or higher | one year

SECONDARY OUTCOMES:
To determine the proportion of subjects whose confirmatory biopsy is upgraded to Gleason score 7 (4 + 3) or higher | one year

CONTACTS AND LOCATIONS:
Overall Officials: Laurence Klotz, MD, Principal Investigator — Canadian Urology Research Consortium
Locations (3):
- Canada (3):
  - London Health Sciences Centre, London, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Princess Margaret Hospital, Toronto, Ontario

REFERENCES:
- [Derived] Klotz L, Pond G, Loblaw A, Sugar L, Moussa M, Berman D, Van der Kwast T, Vesprini D, Milot L, Kebabdjian M, Fleshner N, Ghai S, Chin J, Haider M. Randomized Study of Systematic Biopsy Versus Magnetic Resonance Imaging and Targeted and Systematic Biopsy in Men on Active Surveillance (ASIST): 2-year Postbiopsy Follow-up. Eur Urol. 2020 Mar;77(3):311-317. doi: 10.1016/j.eururo.2019.10.007. Epub 2019 Nov 8. PMID 31708295
- [Derived] Klotz L, Loblaw A, Sugar L, Moussa M, Berman DM, Van der Kwast T, Vesprini D, Milot L, Kebabdjian M, Fleshner N, Ghai S, Chin J, Pond GR, Haider M. Active Surveillance Magnetic Resonance Imaging Study (ASIST): Results of a Randomized Multicenter Prospective Trial. Eur Urol. 2019 Feb;75(2):300-309. doi: 10.1016/j.eururo.2018.06.025. Epub 2018 Jul 13. PMID 30017404